CLINICAL TRIAL: NCT07030582
Title: Efficacy of Internet-Based Cognitive Behavioral Therapy for Back Muscle Strength Loss, Chronic Pain, and Poor Patient Recovery Perceptions After Lumbar Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiawei Jiang (Other)
Responsible Party: Sponsor-Investigator, Jiawei Jiang, Attending Physician, Affiliated 2 Hospital of Nantong University
Organization: Affiliated 2 Hospital of Nantong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TWang
Record Dates: First submitted 2025-05-17; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Internet-Based Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The research team developed a comprehensive core muscle training protocol based on internet-delivered cognitive behavioral therapy through the digital rehabilitation platform.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy; Behavioral: Basic Postoperative Care
- The control group (Active Comparator): The control group received conventional postoperative care interventions
  Interventions: Behavioral: Basic Postoperative Care; Behavioral: Conventional Postoperative Care

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy — The intervention group received a comprehensive core muscle training protocol delivered through a digital rehabilitation platform from hospital admission to 6 months post-surgery. The protocol began with initial screening, including online assessments of cognitive misconceptions, kinesiophobia, and posture analysis. Pain-related cognitive restructuring was addressed through virtual reality sessions, educational videos, and mindfulness breathing guidance. Behavioral activation incorporated graded exposure therapy with EMG biofeedback, interactive knowledge quizzes, and peer modeling. Exercise skills were developed through personalized progressive training with real-time video guidance, and protocols were adjusted based on mid-term assessments. Behavioral reinforcement strategies included recovery support groups, compliance tracking, and integration of exercises into daily activities. A three-tier warning system (Red/Yellow/Green) was implemented to monitor safety and compliance, trigger
  Arms: The intervention group
Behavioral: Basic Postoperative Care — All participants were instructed to maintain their usual daily activities and abstain from additional treatments throughout the 6-month study period.
Behavioral: Conventional Postoperative Care — The control group received conventional postoperative care, which included the establishment of a WeChat support group and provision of a rehabilitation manual focusing on core muscle training on the first postoperative day. Physical therapists provided individualized bedside instruction to ensure proper exercise techniques. Structured follow-up was conducted via telephone or social media (weekly during the first month, then monthly from months 2-6, with each session lasting at least 15 minutes) to provide psychological support and exercise guidance through relaxation techniques and individualized core muscle training progression.
  Arms: The control group

SUMMARY:
This study aims to develop an Internet-based Cognitive Behavioral Therapy protocol for core muscle training, based on an understanding of factors impeding postoperative core muscle training in lumbar surgery patients. The protocol is designed to reconstruct patients' cognition, eliminate adverse behaviors, and promote healthy behaviors such as core muscle training among LDH patients. The ultimate objectives are to alleviate postoperative pain, enhance lumbar stability, and facilitate disease rehabilitation in patients following lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years
* diagnosis of lumbar disc herniation requiring single-level lumbar fusion surgery - no previous history of lumbar surgery
* Surgical procedures performed by the same surgical team
* willingness to comply with the study protocol and restrictions
* availability of a home WiFi connection

Exclusion Criteria:

* lumbar surgery secondary to neoplasm, tuberculosis, infection, or inflammation
* postoperative infection or revision surgery
* presence of cauda equina syndrome
* diagnosis of schizophrenia, cognitive impairment, or other psychiatric disorders
* coexisting severe cardiovascular or cerebrovascular diseases, or congenital conditions precluding exercise participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
TSK Scores | The TSK scores were collected at baseline and at 1 week, 1 month, 3 months, and 6 months post-intervention.
  The Tampa Scale of Kinesiophobia (TSK) was administered to evaluate kinesiophobia in both groups before and after intervention. The TSK is a validated 17-item questionnaire, with each item scored on a 4-point scale. The TSK consists of 17 items with a total score ranging from 17 to 68 points, with higher scores indicating greater severity of kinesiophobia.
Exercise Adherence | Exercise adherence scores were collected at baseline and at follow-up intervals of 1 week, 1 month, 3 months, and 6 months post-intervention.
  The Orthopedic Patient Exercise Compliance Scale total score (ranging from 15 to 75 points) will be used to evaluate patients' adherence to postoperative functional exercises, using a 15-item questionnaire that assesses three dimensions (physical, psychological, and active learning aspects). Each item is scored on a 5-point Likert scale (1 = completely unable to 5 = completely able), with higher total scores indicating better exercise compliance (>55 points represents high adherence, 20-55 points indicates partial adherence, and <20 points indicates low adherence).
Pain Intensit | Pain scores were collected at baseline and follow-up intervals of 1 week (at discharge), 1 month, 3 months, and 6 months post-intervention.
  Pain severity will be measured using the Numerical Rating Scale (NRS) total score (ranging from 0 to 10 points), a validated 11-point scale for pain assessment. Pain levels are categorized according to the following scoring criteria: 0 = no pain, 1-3 points = mild pain, 4-6 points = moderate pain, 7-9 points = severe pain, and 10 points = extreme pain, with higher scores indicating greater pain severity.

SECONDARY OUTCOMES:
Lumbar Function | The JOA scores were collected at baseline, 3 months, and 6 months post-intervention.
  Lumbar functional status will be measured using the Japanese Orthopaedic Association (JOA) scale total score (ranging from 0 to 29 points), a comprehensive assessment tool that evaluates four functional domains: subjective symptoms (low back pain, leg pain, and gait), clinical signs (straight leg raising, sensory disturbance, and motor dysfunction), restriction of activities of daily living, and bladder function, with lower scores indicating more severe functional impairment
Trunk Shift (Spinal Alignment) | Measurements were obtained at baseline, 3 months, and 6 months post-intervention.
  Lateral deviation of vertebra prominens from the midline will be measured using the DIERS FORMETRIC III 4D motion analysis system (DICMA V2.x.x software, DIERS Medical Systems, Beijing, China). The measurement is expressed in millimeters (mm), with larger values indicating greater lateral deviation.
Pelvic Torsion | Measurements will be obtained at baseline, 3 months, and 6 months post-intervention.
  Rotational angle between posterior superior iliac spines will be measured using the same DIERS FORMETRIC III 4D system. The measurement is expressed in degrees (°), with larger values indicating greater pelvic rotation.
Maximum Vertebral Rotation | Measurements will be obtained at baseline, 3 months, and 6 months post-intervention.
  The sum of maximum vertebral rotation angles will be measured using the same DIERS FORMETRIC III 4D system. The measurement is expressed in degrees (°), with larger values indicating greater vertebral rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated 2 Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No